CLINICAL TRIAL: NCT03645629
Title: Comparison of Skin Prick Tests and Atopy Patch Test Results of Lyophilized Food Extracts at Different Storage Time (0, 3 and 6 Months) After Preparation
Brief Title: Efficacy of Lyophilized Food Extracts for Skin Prick Tests and Atopy Patch Test at Different Storage Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 619/2556 (EC 3)
Record Dates: First submitted 2018-08-17; First posted 2018-08-24 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Skin Tests

STUDY DESIGN:
Intervention Model Description: Perform skin prick test and atopy patch test of lyophilized foods (cow milk, egg white, egg yolk, wheat, soy and shrimp) stored at different time; 0, 3 and 6 months after preparation.
  Then compare the results.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Food skin tests at 0 month (Active Comparator): the skin test results of food extract at time 0 months after preparation
  Interventions: Diagnostic Test: skin test with food at different storage times
- Food skin tests at 3 month (Active Comparator): the skin test results of food extract at time 3 months after preparation
  Interventions: Diagnostic Test: skin test with food at different storage times
- Food skin tests at 6 month (Active Comparator): the skin test results of food extract at time 6 months after preparation
  Interventions: Diagnostic Test: skin test with food at different storage times

INTERVENTIONS:
Diagnostic Test: skin test with food at different storage times — Perform skin tests to each foods at 0, 3, 6 months after preparation and compare the results

SUMMARY:
Comparison the result of skin prick tests and atopy patch test of lyophilized food extracts at different storage time (0, 3 and 6 months) after preparation

DETAILED DESCRIPTION:
Skin prick test were performed with lyophilized food extracts (cow milk, egg white, egg yolk, wheat, soy and shrimp) at different storage time (0, 3 and 6 months) after preparation.

Atopy patch test were performed with lyophilized food extracts (cow milk, egg white, egg yolk, wheat, soy and shrimp) at different storage time (0, 3 and 6 months) after preparation

ELIGIBILITY:
Inclusion Criteria:

* mild to moderately severe food allergy patients
* At least positive skin test to one kind of common food (commercial extract)
* Stop antihistamine or corticosteroid (if more than 20mg/day) for at least 7 days

Exclusion Criteria:

* Dermographism
* Severe systemic disease such as autoimmune disease, immune deficiency, malignancy
* Severe dermatitis or large area involment
* pregnancy

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
skin test result of lyophilized foods at 6 months after preparation | 6 month
  Perform skin prick test and atopy patch test the patients with lyophilized foods at 0, 3 and 6 months after preparation and compare the results at 6 months to 0 and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nualanong Visitsunthorn, MD, Principal Investigator — Department of Pediatrics, Siriraj hospital, Mahidol University
Locations (1):
- Siriraj Hospital. Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Publication